CLINICAL TRIAL: NCT04981275
Title: A Multi-omic Approach to Evaluate and Characterize the Polycystic Ovary Syndrome (PCOS) Phenotype
Status: Completed | Type: Observational
Sponsor: Onegevity Health (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Other Study IDs: HP-00089723
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, saliva, vaginal microbiome, stool microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with PCOS: Women previously diagnosed with PCOS not using hormonal therapy and without other significant health or endocrine issues
  Interventions: Other: No intervention study
- Healthy controls: Women self-identifying as generally healthy, not using hormonal therapy, and without any significant health or endocrine issues
  Interventions: Other: No intervention study

INTERVENTIONS:
Other: No intervention study — This observational study will only collect data, not provide any intervention to participants.

SUMMARY:
The purpose of this research study is to explore the relationship between the gut microbiome and hormone levels in women diagnosed with PCOS and determine whether there are differences in the gut microbiome between women with PCOS and women without PCOS.

Consented, enrolled participants will complete a health questionnaire, complete a fasted blood draw at a local laboratory, and provide a stool, saliva, and vaginal swab sample for comprehensive biomarkers, hormones, metagenomics, and metabolomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS or Women who are considered Healthy
* 18-40 years old
* Residing in the USA, except for exclusion states
* Have not been using hormonal therapy for at least 3 months

Exclusion Criteria:

* Women using hormonal therapy within the last 3 months
* Diagnosed with other significant health conditions or using medications that will affect hormone levels
* Residing in NY, NJ, MD, RI, ND, SD, or HI
* Pregnant or nursing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, ages 18-40, living in the USA (except for NY, NJ, RI, MD, SD, ND, or HI), who have not been using hormonal therapy for at least 3 months and without other significant health issues or medications affecting hormones. Women must be previously diagnosed with PCOS or considered Healthy and not currently pregnant or nursing. Women will be referred to the study by their Physician or word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Phenotype differences in vaginal microbiome | Samples to be collected on any day once per participant within 30 days of enrollment
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Vaginal swabs are to be collected by women and analyzed with metagenomics and metabolomics sequencing.
Phenotype differences in gut microbiome | Samples to be collected once on any day per participant within 30 days of enrollment
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Stool samples are to be collected by women and analyzed with metagenomics sequencing.
Phenotype differences in blood biomarkers | Samples to be collected once within a 5-day window to control for menstrual cycle, within 30 days of enrollment
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Venipuncture blood draws are to be completed and analyzed by a commercial laboratory, for a comprehensive analysis of targeted hormones and untargeted metabolic systems.
Phenotype differences in DNA | Samples to be collected once per participant within 30 days of enrollment
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Saliva samples are to be collected and analyzed by a commercial laboratory for DNA and metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Chris D'Adamo, PhD, Principal Investigator — University of Maryland; Chris Mason, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided